CLINICAL TRIAL: NCT03259633
Title: An Intermediate Access Protocol for Selumetinib for Treatment of Neurofibromatosis Type 1 With Inoperable, Progressive/Symptomatic Plexiform Neurofibromas (PN)
Brief Title: An Intermediate Access Protocol for Selumetinib for Treatment of Neurofibromatosis Type 1
Status: Approved for marketing | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1346R00002; D1346R00002 (Other: Astra Zeneca)
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: NF type1 With Inoperable Plexiform Neurofibromas
Keywords: Neurofibromatosis type1,; Plexiform Neurofibromas; inoperable, progressive/symptomatic plexiform neurofibromas (PN) without any alternative therapeutic options; mutation in the NF1 gene; Selumetinib; Early Access; Intermediate Access Protocol
MeSH Terms: conditions — Neurofibroma, Plexiform | interventions — AZD 6244

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Selumetinib — open-label, single-arm, multicenter intermediate access protocol

SUMMARY:
This will be an open-label, single-arm, multicenter intermediate access protocol which provides treatment access to selumetinib for eligible patients with neurofibromatosis type 1 (NF1) who have inoperable, progressive/symptomatic plexiform neurofibromas (PN) without any alternative therapeutic options. All patients will continue to receive drug while they are deriving clinical benefit.

Approximately 100 patients in the US will be treated as part of this protocol

DETAILED DESCRIPTION:
Patients must have received a clinical diagnosis of NF1 and have inoperable, progressive/symptomatic PN, where inoperable is defined as PN that cannot be surgically completely removed without risk of substantial morbidity.

The population are patients with NF1 who have inoperable, progressive/symptomatic PN aged ≥ 2years with onset of disease before they were 18 years and who have demonstrated an ability to swallow whole capsules, who have no further treatment options and are not eligible for clinical trials.

There is no maximum duration for selumetinib treatment. Patients may continue to receive selumetinib as long as they continue to show clinical benefit, as judged by the treating physician, and in the absence of unacceptable toxicity.

Once patients have been discontinued from treatment, other available treatment options will be at the discretion of the physician

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of neurofibromatosis type 1 (NF1) and have inoperable, progressive/symptomatic plexiform neurofibromas (PN)
2. Presence of inoperable PN , defined as a PN that cannot be surgically completely removed without risk for substantial morbidity
3. Patients aged ≥2 with onset of disease before they were 18 years and a BSA ≥ 0.55 m2 who are able to swallow whole capsules. (approx. length 15.4 mm, diameter 5.4 mm). A swallow test must be performed before requesting drug
4. Normal cardiac function defined as normal ejection fraction (ECHO, MUGA or cardiac MRI) as per institutional normal and absence of prior heart disease
5. Adequate blood pressure as defined in line with local practice.
6. The patient has exhausted all available approved therapies as appropriate for NF1 with inoperable progressive/symptomatic PN
7. Provision of a signed informed consent prior to any protocol specific procedures. Patients already receiving selumetinib through single patient access who enroll in this protocol must be reconsented and sign the consent form for this intermediate access protocol.
8. For female patients of childbearing potential, have evidence of a post-menopausal status, or a negative urinary or serum pregnancy test.

Exclusion Criteria:

1. Unresolved chronic toxicity ≥ CTCAE Grade 2 from previous therapy
2. Patients eligible for any ongoing clinical trials with selumetinib in the indication in question
3. Ophthalmological conditions: Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR) or retinal vein occlusion Intraocular pressure (IOP) should not be > 21 mmHg for adults or outside the range of normal for children or uncontrolled glaucoma (irrespective of IOP)
4. Male or female patients of reproductive potential and, as judged by the investigator, are not employing an effective method of birth control.
5. Female patients who are breast-feeding.
6. Have evidence of any other significant clinical disorder or laboratory finding that, as judged by the treating physician, makes it undesirable for the patient to participate in the study.
7. Have any evidence of a severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease, active infection (including hepatitis B, hepatitis C, HIV), active bleeding diatheses or renal transplant
8. Have refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would adversely affect the absorption / bioavailability of the orally administered study medication

Ages: 2 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Bornhorst, MD, Principal Investigator — Investigator
Locations (1):
- Research Site, New Orleans, Louisiana, United States